CLINICAL TRIAL: NCT06464731
Title: Endovascular Treatment for Mild Ischemic Stroke Due to Acute Large Vessel Occlusion in the Anterior Circulation: A Multicenter Prospective Registry
Brief Title: Endovascular Treatment for Mild Ischemic Stroke Due to Acute Large Vessel Occlusion in the Anterior Circulation
Acronym: Mild-MT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wen-huo Chen (Other)
Responsible Party: Sponsor-Investigator, Wen-huo Chen, Professor, Zhangzhou Municipal Hospital
Organization: Zhangzhou Municipal Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mild-MT registry
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Endovascular Treatment; Mild Stroke
Keywords: endovascular treatment; mild stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The operator will choose the optimal endovascular treatment strategy and device based on the patient's condition and clinical experience. This may include, but is not limited to, stent retriever thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, balloon angioplasty, stent implantation, etc. The endovascular treatment plan and relevant time points will be accurately recorded. The patient will receive the best medical treatment according to current local clinical research standards during and after the procedure.
  Interventions: Procedure: EVT
- Control Group (No Intervention): Patients will receive the best medical treatment according to local clinical research standards, including antiplatelet agents, anticoagulants, thrombolysis, etc., excluding any endovascular treatment. In the event of disease progression defined as neurological deterioration leading to an increase in NIHSS ≥4 points and excluding non-stroke factors within 24 hours, remedial endovascular treatment may be taken, including but not limited to stent retriever thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, balloon angioplasty, stent implantation, etc.

INTERVENTIONS:
Procedure: EVT — Interventionist choose the optimal EVT strategy and device based on the patient's condition and local guidelines. This may include, but not limited to, stent-retriever thrombectomy, aspiration thrombectomy, intra-arterial thrombolysis, balloon angioplasty, stent implantation and so on. The EVT regimen and relevant time points will be accurately recorded. The patient will receive the best medical treatment according to the local guidelines.
  Other Names: Experimental
  Arms: Experimental Group

SUMMARY:
Explore the effectiveness and safety of emergency endovascular treatment in patients with mild ischemic stroke due to acute large vessel occlusion in the anterior circulation, identified through perfusion imaging.

DETAILED DESCRIPTION:
The purpose of this registry is to select patients with mild AIS caused by anterior circulation LVO with mismatched volume of the ischemic penumbra based on screen of cerebral perfusion imaging. This registry aim to explore the efficacy and safety of EVT for mild AIS patients with anterior circulation large vessel occlusion within 24 hours of onset.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Symptoms onset or last known well to randomization is within 24 hours.
3. Clinical diagnosis of acute ischemic stroke due to anterior circulation intracranial large vessel occlusion (LVO) (including intracranial internal carotid artery [ICA], middle cerebral artery [MCA] M1 segment, MCA M2 segment, with or without ipsilateral extracranial ICA occlusion) confirmed on Computerized tomography angiography (CTA) or Magnetic resonance imaging angiography (MRA) ;
4. Baseline NIHSS score <6 before randomization (including cases with NIHSS ≥6 at onset but improves before randomization);
5. ASPECTS score ≥6 based on Non-contrast CT (NCCT) before randomization;

Exclusion Criteria:

1. Premorbid Rankin Scale (mRS) score ≥ 1;
2. Known allergy to iodine, heparin, anaesthesia, or other definite contraindication to receiving endovascular treatment (EVT) procedure;
3. Patient has severe or fatal co-morbidities that could interfere with outcome assessments and follow-up (such as malignant tumor, severe heart failure, or renal failure, or life expectancy less than 6 months);
4. Poorly controlled hypertension (systolic blood pressure >220 mmHg or diastolic blood pressure >120 mmHg);
5. Baseline blood glucose <50mg/dL (2.78 mmol/L) or >400mg/dL (22.20 mmol/L);
6. Known bleeding tendencies, including but not limited to platelet count <100×109/L; received heparin treatment within 48 hours with an activated partial thromboplastin time (APTT) ≥35s; recent oral anticoagulant therapy with international normalized ratio (INR) >3; Note: Patients without a history of coagulation abnormalities or without suspicion of coagulation abnormalities do not need to wait for laboratory test results before enrollment;
7. Seizures at stroke onset or during the course, hard to accurately judge the baseline NIHSS score;
8. Female who is known to be pregnant, lactation, or tested positive for pregnancy at time of admission;
9. Currently participating in another investigational drug study or medical device treatments that may interfere with the results of this study;
10. Evidence of intracranial hemorrhage on CT/MRI, including cerebral parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, and subdural/extradural hemorrhage;
11. Significant midline displacement, hernia of brain, or ventricular mass effect with midline displacement confirmed on CT/MRI;
12. Anticipated impossibility to complete endovascular treatment, such as vascular tortuosity, severe vascular wall calcification, etc.;
13. Aortic dissection;
14. Multiple intracranial large vessel occlusions confirmed by CTA or MRA, unable to clearly identify the symptomatic vessel, such as bilateral MCA occlusions or occlusions involving both the MCA and basilar artery;
15. Suspected or confirmed occluded artery is non-acute occlusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-09-11 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The rate of excellent outcome | 90±7 days
  mRS score 0-1

SECONDARY OUTCOMES:
The rate of good outcome | 90±7 days
  mRS score 0-2
mRS shift | 90±7 days
  distribution of mRS scores

OTHER OUTCOMES:
The rate of symptomatic intracranial hemorrhage | Within 48 hours
  According to the Heidelberg criteria
Rate of early neurological deterioration | Within 7 days
  An increase in NIHSS≥4 or an increase of ≥2 in any individual item
Mortality | 90±7 days
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Tingyu Yi, MD, Principal Investigator — Zhangzhou Affiliated Hospital
Locations (9):
- China (9):
  - Zhangzhou Municipal Hospital, Zhangzhou, Fujian
  - Gansu Provincial Hospital of Traditional Chinese Medicine, Lanzhou, Gansu
  - Jiamusi Central Hospital, Jiamusi, Heilongjiang
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Songyuan Jilin Oilfield Hospital, Songyuan, Jilin
  - Shenyang First People's Hospital, Shenyang, Liaoling
  - Lishui Central Hospital, Lishui, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No